CLINICAL TRIAL: NCT05891314
Title: The Effect of Botulinum Toxin Injection After Hemorrhoidectomy in Pain Control: a Randomized Controlled Trial
Brief Title: The Effect of Botulinum Toxin Injection After Hemorrhoidectomy in Pain Control.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmad Sakr, consultant and lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5678
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Pain; Haemorriodectomy; Anal Sphincterotomy
Keywords: post hemorridectomy pain; sphincterotomy; botox injection
MeSH Terms: conditions — Pain | interventions — Lateral Internal Sphincterotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botox injection post hemorridectomy (Active Comparator): after piles excision this group will be subjected to botox injection in the internal sphincter
  Interventions: Procedure: Botox Injectable Product; Procedure: Internal sphincterotomy
- Hemorridectomy alone (No Intervention): Just hemorridectomy without botox injection(control group)
- Hemorridectomy plus internal sphincterotomy (Active Comparator): after piles excision patients will undergo internal sphincterotomy
  Interventions: Procedure: Botox Injectable Product; Procedure: Internal sphincterotomy

INTERVENTIONS:
Procedure: Botox Injectable Product — one group will have botox injection in the internal sphincter
  Other Names: Botulonium toxin injection
  Arms: Botox injection post hemorridectomy; Hemorridectomy plus internal sphincterotomy
Procedure: Internal sphincterotomy — this group will have internal sphincterotomy
  Other Names: lateral internal sphincterotomy
  Arms: Botox injection post hemorridectomy; Hemorridectomy plus internal sphincterotomy

SUMMARY:
Hemorrhoids are a common disease in the general population. Its prevalence is estimated to be 5-36 % and more prevalent in western countries . Half of people older than 50 years of age will suffer from hemorrhoids in a period of their life, of which only 5-10% will require surgical intervention while most of the remainders become asymptomatic and improved with the conservative treatment.

Conservative treatment in the form of diet modification as well as some medical treatment, is usually effective. On the other hand, a few patients require surgical intervention. Surgery is indicated for those not responding to conservative management, those with grade III, and grade IV hemorrhoids.

Surgical treatment is the only curative method for hemorrhoidal disease and indicated for advanced and complicated disease. The most radical operations with the best results are the Milligan-Morgan and Ferguson hemorrhoidectomy .

However, the major concern of hemorrhoidectomy is the post-operative pain that occurs in 20-40 % of patients and it is considered the main cause of refusing surgery. The cause of postoperative pain is multifactorial, including the type of anesthesia , hemorrhoidectomy technique. and spasm of the internal anal sphincter (IAS) that becomes exposed after hemorrhoidectomy. The spasm of the IAS is considered the target to relieve pain post operatively. Lateral internal sphincterotomy (LIS) is widely used as an adjunct to relieve pain post hemorrhoidectomy as it release the spasm of the sphincter and subsequently relieve pain. However, this procedure is not accepted by many surgeons due to its recorded complications as bleeding and mild degree of fecal incontinence, so its role following hemorrhoidectomy is still controversial.

On the other hand, the spasm of the anal sphincter can be abolished by injection of the botulinum toxin which acts on the acetylcholine receptor and consequently temporary muscle paralysis occurs that is followed by decreased pain and wound healing.

Our hypothesis is botulinum toxin relaxes the internal sphincter, so prevent its spasm and so reducing the pain and promoting wound healing more rapidly.

DETAILED DESCRIPTION:
many procedures have been described to decrease the pain post hemorridectomy. Internal sphincterotomy Botox Injection giving strong analgesics

We aim to evaluate the efficacy of Botox and internal sphincterotomy in pain relief after hemorridectomy.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes,
* aged between 18 and 70 years old.
* Grade III and IV hemorrhoids.
* Those with failed conservative treatment.

Exclusion Criteria:

* surgically unfit patients due to multiple comorbidities,
* patients who need emergency operation for complicated hemorrhoids,
* patients with partial rectal prolapse
* patients with rectal varices due to portal hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 2weeks
  according to the visual analogue scale (VAS), which contain 10 degrees, the lower the degree , the lower the score this means less pain.

SECONDARY OUTCOMES:
Time taken to return to daily activities in days. | 4-6weeks
  return to daily activities without complaint

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad, Al Mansurah, Egypt